CLINICAL TRIAL: NCT06597604
Title: Evaluation of the Effectiveness and Security of TenaTac® in the Prevention of Air Leaks in Thoracic Surgery
Acronym: TENATAC
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hopitaux Prives de Metz, Groupe UNEOS (Other)
Collaborators: CuraMedrix B.V. (Unknown); Medical Advices Consulting (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PI-2024-002; 2024-A01716-41 (Other: ID-RCB)
Record Dates: First submitted 2024-09-12; First posted 2024-09-19 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Lung Surgery
Keywords: Lung surgery; TenaTac; Gelatin Patch; Sealant; PAL; Pulmonary Air Leak; Lobectomy
MeSH Terms: interventions — Pulmonary Surgical Procedures

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental Group (Experimental): Thoracic Surgeons will apply the experimental device TenaTac® after major lung resection
  Interventions: Device: Intraoperative use of TenaTac in lung surgery
- Control Group (Active Comparator): Thoracic Surgeons will apply other (usual) sealing device after major lung resection
  Interventions: Device: Intraoperative use of usual sealant in lung surgery

INTERVENTIONS:
Device: Intraoperative use of TenaTac in lung surgery — Use of innovative medical device : TenaTac
  Arms: Experimental Group
Device: Intraoperative use of usual sealant in lung surgery — Use of the usual scealant as a control
  Arms: Control Group

SUMMARY:
Lung surgery remains a high-risk procedure, with serious adverse events that can occur later, including postoperative bleeding or hemothorax, pneumopathy or surgical site infection but also ... per- and post-operative air leaks. Majority the air leaks resolve spontaneously within 48 hours but certain cases persist within several days which known as prolonged air leaks, or PAL. Several safe and effective sealing agents are used to contain and or reduce the intensity and incidence of postoperative air leaks, and the time required for drain removal. This protocol assesses the effectiveness of an innovative gelatin-based medical device named TenaTac® (Selentus Science, UK) in preventing air leak after major lung resection.

DETAILED DESCRIPTION:
Thoracic surgery is a specialty dedicated to the management (diagnosis and treatment...) of conditions and lesions of the thoracic cage and its organs, excluding the heart, aorta and esophagus. It is based on 2 surgical techniques: open (by posterolateral thoracotomy) or minimally invasive endoscopic (with or without robot-assisted surgery).

Lobectomy is the most common pulmonary resection, however, regardless of the surgical option chosen, lung surgery remains a high-risk procedure, with serious adverse events that can occur later, including postoperative bleeding or hemothorax, pneumopathy or surgical site infection, pulmonary alveolar collapse, acute respiratory distress syndrome, pleural or pericardial effusion, lobar torsion or multi-organ failure, bronchial or esophageal fistulas, transient arrhythmia due to vagus nerve damage, pulmonary embolism, venous ischemia, ... and, per- and post-operative air leaks. Air leak has been reported in 25-75% of patients, which makes it the most common incident after elective lung surgery.

Although the majority of these air leaks resolve spontaneously within 48 hours (by continuous pleural drainage), certain cases persist for several days (more than 5 days). These are known as prolonged air leaks, or PAL.

The literature describes several sealing agents used to contain air leaks. The preventive use of sealants at the lung resection site seems safe and effective, since it significantly reduces the intensity and incidence of postoperative air leaks, and the time required for drain removal, Pharmaceutical gelatin-based medical devices, used for decades for their hemostatic properties, have recently been suggested for sealing pulmonary defects and preventing air leaks. Regarding the results obtained, gelatin appears to be a therapeutically effective biomaterial in lung surgery. We therefore hypothesize the effectiveness of the innovative medical device TenaTac® (Selentus Science, UK) in preventing air leak after major lung resection.

ELIGIBILITY:
Inclusion Criteria:

* Patients hospitalized in the thoracic surgery departments of the investigating centers, for elective surgery,
* Lobectomy surgery requiring the use of a sealing agent,
* Adult patients (>18 years),
* Patients who have given written consent to participate in the study,
* Patients registered within the social security insurance in France.

Exclusion Criteria:

* Patients hospitalized in emergency,
* Patients with gelatin allergy,
* Patients undergoing other biomedical research likely to interfere with the evaluation criteria of this study
* Patients under tutorship and/or curatorship,
* Patients unable to follow the planned post-operative follow-up,
* Patients whose life expectancy is less than 1 year,
* Pregnant or breast-feeding patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
To compare the effectiveness of the TenaTac® patch on the duration of thoracic drainage for each patient (regardless of their degree of emphysema) compared to sealing devices routinely used by thoracic surgeons for the same indication | 4 weeks
  Assess the effectiveness of the TenaTac® patch in terms of duration of thoracic drainage, compared with sealing devices routinely used by thoracic surgeons for the same indication.

SECONDARY OUTCOMES:
To assess the effectiveness of the TenaTac® patch in preventing postoperative air leaks throughout the hospital stay, and more specifically in PALs (beyond the 5th day). | 4 weeks
  Assess the effectiveness of the TenaTac® patch in terms of PAL rates decrease compared to those measured with the other sealants routinely used by thoracic surgeons for the same indication and in the same circumstances
Effectiveness of the TenaTac® patch in reducing hospital stay | 4 weeks
  Assess the effectiveness of the TenaTac® patch in reducing hospital stay, compared to those obtained with the other sealants routinely used by thoracic surgeons for the same indication and in the same circumstances
Effectiveness of the TenaTac® patch in preventing (immediate and medium term) postoperative complications | 4 weeks
  Assess the effectiveness of the TenaTac® patch in preventing (immediate and medium term) postoperative complications, compared to those declared with the other sealants routinely used by thoracic surgeons for the same indication and in the same circumstances

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro ORSINI, MD, Principal Investigator — Hôpitaux Privés de Metz, Groupe UNEOS
Locations (2):
- France (2):
  - Hôpital Robert Schuman_Groupe UNEOS, Metz, Grand Est
  - Centre Hospitalier de la Côte Basque (Bayonne), Bayonne

IPD SHARING:
Plan to Share IPD: Yes
Data collected throughout the trial used in the results publication will be shared with other researchers